CLINICAL TRIAL: NCT05745454
Title: A Phase I Clinical Study on the Safety and Efficacy of Chimeric Antigen Receptor T-cell (CART) in the Treatment of Human Epidermalgrowth Factor Receptor-2 (HER2) Positive and Refractory Advanced Solid Tumors
Brief Title: A Clinical Study on the Safety and Efficacy of Chimeric Antigen Receptor T-cell (CART) in the Treatment of Solid Tumors
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: su haichuan (Other)
Responsible Party: Sponsor-Investigator, su haichuan, Head of Department, Tang-Du Hospital
Organization: Tang-Du Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HER2-E-CART
Record Dates: First submitted 2022-12-08; First posted 2023-02-27 (Actual); Last update posted 2023-02-27 (Actual); Status verified 2023-02

CONDITIONS: Solid Tumor

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HER2-E-CART cells (Experimental): HER2-E-CART cells were intravenously transfused and followed up to 2 years after the last cell transfusion
  Interventions: Biological: HER2-E-CART cells

INTERVENTIONS:
Biological: HER2-E-CART cells — E-CAR-T is a novel second-generation CAR-T product targeting HER2 protein

SUMMARY:
This is a single-arm, investigator-initiated exploratory study.The study is designed to evaluate the safety and the tolerability of HER2-E-CART cells for the treatment of patients with HER2-positive, refractory advanced solid tumors in three dose groups: low, medium and high.

DETAILED DESCRIPTION:
This study was a one-arm,investigator-initiated exploratory study. According to the "3+3" principle, three dose groups with increasing dose were set up, namely low, medium and high dose groups, with separate cell counts. A total of 9-12 subjects were enrolled in the group and given intravenous infusion. Dose-limited toxicity was observed from the beginning of preconditioning to 28 days after CAR T infusion.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily signed an informed consent form and were able to complete the study procedures and follow-up examinations and treatment
2. Age ≥ 18 years and ≤ 70 years, regardless of gender
3. Weight > 40 kg
4. Eastern Cooperative Oncology Group (ECOG) physical status score of 0 to 1
5. Patients with refractory advanced solid tumors who have failed or are intolerant of existing standard regimens or whose patients have refused standard regimens
6. The presence of at least one measurable lesion according to Response Evaluation Criteria In Solid Tumors 1.1 criteria
7. With good organ function
8. Positive HER2 cell membrane expression
9. Women of childbearing potential must have a pregnancy test with negative results within 7 days prior to initiation of treatment

Exclusion Criteria:

1. Any systemic antitumor therapy within 2 weeks prior to the single blood collection
2. History of organ transplantation
3. Pregnant or lactating women
4. Uncontrolled infectious disease, such as baseline Hepatitis B Virus DNA ≥ 1000 IU/ml, anti-HIV positive, Hepatitis C Virus-RNA positive
5. Other clinically significant active infections
6. Other active malignancies within the previous 5 years, such as basal or squamous skin cancer, superficial bladder cancer, or in situ breast cancer that has been completely cured and does not require follow-up treatment subjects are not included
7. Patients with severe autoimmune or immunodeficiency diseases, such as subjects with a confirmed diagnosis of a severe autoimmune disease requiring systemic immunosuppressive (steroid) therapy for a prolonged period of time (more than 2 months) or with immune-mediated symptomatic diseases, including ulcerative colitis, Crohn's disease, rheumatoid arthritis, systemic lupus erythematosus (SLE), autoimmune vasculitis (e.g., Wegener's granulomatosis), etc
8. Subjects with known severe allergic reactions to pretreatment drugs such as injectable cyclophosphamide, injectable paclitaxel (albumin-bound), or CAR-T cell preparations including adjuvants, dimethylsulfoxide
9. Any unstable systemic disease: including but not limited to unstable angina pectoris, cerebrovascular accident or transient ischemia (within 6 months prior to screening), myocardial infarction (within 6 months prior to screening), New York Heart Association (NYHA) classification ≥ Class III congestive heart failure, severe arrhythmias poorly controlled by medications, liver, kidney or metabolic disease, and hypertension uncontrolled by standard therapy 10
10. Those with active bleeding, thrombotic disorders requiring treatment
11. Patients with pericardial, thoracic, or abdominal effusions requiring clinical management or intervention
12. The presence of known or suspected brain metastases, including central nervous system and spinal cord compressions or meningeal metastases
13. Subjects undergoing treatment with systemic steroids or steroid inhalers
14. Subjects with any psychiatric disorder, including dementia, altered mental status, that may interfere with informed consent and understanding of relevant questionnaires
15. Having participated in another clinical trial within the previous 30 days
16. Have received a live or attenuated vaccine within 4 weeks prior to pretreatment
17. Those who have been judged by the investigator to have a serious uncontrollable disease or have other conditions that may interfere with receiving treatment in this study and are considered unsuitable

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2023-02 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Occurence of Adverse event rate | Adverse events will be collected from the beginning to the end of the study, up to 2 years after the last cell transfusion
  The occurrence of all adverse events (AEs), serious adverse events (SAEs) and treatment-related adverse events (TEAEs).

SECONDARY OUTCOMES:
Time to peak of serum cytokine Interleukin-2 | Within 72 hours before lymphodepletion pretreatment, within 24 hours before and 1 hour after reinfusion, 24 hours, Day 4, Day 7, Day 10, Day 14, Day 28, Day 60, Day 90, Day 180, Day 270, Day 360.
  Time to peak of serum cytokine Interleukin-2
Time to peak of serum cytokine Interleukin-6 | Within 72 hours before lymphodepletion pretreatment, within 24 hours before and 1 hour after reinfusion, 24 hours, Day 4, Day 7, Day 10, Day 14, Day 28, Day 60, Day 90, Day 180, Day 270, Day 360.
  Time to peak of serum cytokine Interleukin-6
Time to peak of serum cytokine Interleukin-10 | Within 72 hours before lymphodepletion pretreatment, within 24 hours before and 1 hour after reinfusion, 24 hours, Day 4, Day 7, Day 10, Day 14, Day 28, Day 60, Day 90, Day 180, Day 270, Day 360.
  Time to peak of serum cytokine Interleukin-10
Time to peak of serum cytokine Tumor Necrosis Factor-α | Within 72 hours before lymphodepletion pretreatment, within 24 hours before and 1 hour after reinfusion, 24 hours, Day 4, Day 7, Day 10, Day 14, Day 28, Day 60, Day 90, Day 180, Day 270, Day 360.
  Time to peak of serum cytokine Tumor Necrosis Factor-α
Time to peak of serum cytokine Tumor Necrosis Factor-γ | Within 72 hours before lymphodepletion pretreatment, within 24 hours before and 1 hour after reinfusion, 24 hours, Day 4, Day 7, Day 10, Day 14, Day 28, Day 60, Day 90, Day 180, Day 270, Day 360.
  Time to peak of serum cytokine Tumor Necrosis Factor-γ
Overall survival (OS) | Baseline up to death event.
  From randomization to the time of death from any cause
Objective Response Rate (ORR) | Baseline up to 144 weeks
  The proportion of patients with tumor size reduction of a predefined amount and for a minimum time period
Disease Control Rate (DCR) | Baseline up to 144 weeks
  The percentage of patients with advanced or metastatic cancer who have achieved complete response (CR), partial response (PR) and stable disease (SD) to a cancer treatment in clinical trials
Duration of Response (DOR) | Baseline up to 144 weeks
  The time from the date of first documentation of a CR or PR or PD to the date of first documentation of tumor progression.
Progression Free Survival (PFS) | Baseline up to 144 weeks
  The time from the first dose to the first documentation of progressive disease (PD) or death from any cause,whichever occurs first
Effects on subjects' health-related quality of life | Baseline up to 144 weeks
  Quality of life related scale ，for questions 1 to 28, choose a number from 1 to 4, 1 means none and 4 means very good. For questions 29 and 30, choose a number from 1 to 7, with 1 being very poor and 7 being very good.
Peak concentration (Cmax) | Within 72 hours before lymphodepletion pretreatment, within 24 hours before and 1 hour after reinfusion, 24 hours, Day 4, Day 7, Day 10, Day 14, Day 28, Day 60, Day 90, Day 180, Day 270, Day 360.
  Maximum plasma drug concentration
Area Under The Curve（AUC） | Within 72 hours before lymphodepletion pretreatment, within 24 hours before and 1 hour after reinfusion, 24 hours, Day 4, Day 7, Day 10, Day 14, Day 28, Day 60, Day 90, Day 180, Day 270, Day 360.
  Area under the plasma concentration-time curve Single dose
Time to Maximum Plasma Concentration（Tmax） | Within 72 hours before lymphodepletion pretreatment, within 24 hours before and 1 hour after reinfusion, 24 hours, Day 4, Day 7, Day 10, Day 14, Day 28, Day 60, Day 90, Day 180, Day 270, Day 360.
  The time required to reach peak concentration after administration
Elimination half-life (t1/2)-Single dose | Within 72 hours before lymphodepletion pretreatment, within 24 hours before and 1 hour after reinfusion, 24 hours, Day 4, Day 7, Day 10, Day 14, Day 28, Day 60, Day 90, Day 180, Day 270, Day 360.
  t1/2 is time it takes for the blood concentration of HER2-E-CART cells or metabolite(s) to drop by half

CONTACTS AND LOCATIONS:
Overall Officials: Haichuan Su, Doctor, Principal Investigator — The Second Affiliated Hospital of PLA Air Force Medical University